CLINICAL TRIAL: NCT05381129
Title: The Effect of Accompanying Temporomandibular Joint Dysfunction on Pain, Quality of Life, Sleep and Functionality in Patients With Chronic Migraine
Brief Title: The Effect of Accompanying Temporomandibular Joint Dysfunction in Patients With Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Alper mengi, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 26.04.2022/373110
Record Dates: First submitted 2022-05-14; First posted 2022-05-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chronic Migraine, Headache; Temporomandibular Joint Dysfunction; Chronic Pain; Quality of Life; Sleep; Headache
MeSH Terms: conditions — Headache; Temporomandibular Joint Disorders; Chronic Pain | interventions — Quality of Life; Sleep; Functional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic migraine (Other): Patients diagnosed with chronic migraine according to the International Headache Society Classification (ICHD-3).
  Interventions: Other: Detection of Pain, Quality of Life, Sleep and Functioning
- Temporomandibular dysfunction (Other): Patients diagnosed with chronic migraine according to the International Headache Society Classification (ICHD-3), and patients with temporomandibular dysfunction.
  Interventions: Other: Detection of Pain, Quality of Life, Sleep and Functioning; Other: Temporomandibular joint dysfunction

INTERVENTIONS:
Other: Detection of Pain, Quality of Life, Sleep and Functioning — All patients will be evaluated for allodynia, quality of life, headache-related disability, and sleep quality.
Other: Temporomandibular joint dysfunction — Patients with jaw complaints will be evaluated for temporomandibular joint dysfunction.
  Arms: Temporomandibular dysfunction

SUMMARY:
The aim of this clinical study to evaluate the effect of temporomandibular joint dysfunction accompanying patients with chronic migraine on pain, quality of life, sleep and functionality.

DETAILED DESCRIPTION:
Patients who applied to Istanbul University - Cerrahpasa, Cerrahpasa Faculty of Medicine, Department of Neurology, headache outpatient clinic and were diagnosed with chronic migraine according to the International Headache Society Classification (ICHD-3), after the patient's history and physical examination, will be included in the study.

Date of birth, gender, education level, body mass index, occupation, marital status, socioeconomic status, age of onset of migraine complaints, descriptive information about migraine attacks (type (with or without aura), duration of attacks, mean number of days with pain) , pain intensity, accompanying) will be questioned.

In addition, patients with complaints and findings such as pain in the temporomandibular joint area and chewing muscles, limitation in mouth opening, noise from the joint during mouth opening and/or non-harmonic jaw movements will be evaluated by Alper Mengi in terms of temporomandibular joint dysfunction.

A total of 62 patients are planned to be included in the study. In the study, 2 groups will be formed, the first group will consist of chronic migraine patients, the second group will consist of patients with chronic migraine as well as temporomandibular joint dysfunction.

All patients will be evaluated for allodynia, quality of life, headache-related disability, and sleep quality. Relevant forms will be filled by patients.

Patients who are thought to have temporomandibular joint dysfunction will be evaluated by Alper Mengi for dysfunction.

ELIGIBILITY:
Inclusion Criteria:

For patients with chronic migraine:

* Being diagnosed with chronic migraine according to the International Headache Society Classification (ICHD-3)
* Being literate

For patients with temporomandibular dysfunction :

* Diagnosed with chronic migraine according to the International Headache Society Classification (ICHD-3)
* Being literate
* Pain in the temporomandibular joint region and chewing muscles for at least 3 months, limitation in mouth opening, noise from the joint when opening the mouth, and / or having complaints and findings such as non-harmonic jaw movements
* Getting a score of ≥1 according to the Helkimo Clinical Craniomandibular Dysfunction Index

Exclusion Criteria:

For patients with chronic migraine:

* Complaint of chronic pain in another part of their body other than the head and face region
* Having another pathology that can explain their pain in the head and face region other than chronic migraine (such as sinusitis, tension-type headache, trigeminal neuralgia, drug overuse headache)
* Psychiatric disease or using psychiatric drugs
* History of serious head trauma or neurosurgical intervention
* Those with a history of infectious, chronic inflammatory disease, malignancy
* Pregnant and breastfeeding women
* History of additional neurological disease other than migraine
* Uncooperative
* Having congestive heart failure, chronic kidney failure, chronic liver disease, lung disease, uncontrolled diabetes, peripheral vascular disease

In addition to the exclusion criteria above in patients with a diagnosis of temporomandibular joint dysfunction:

* Presence of trauma or operation in the temporomandibular joint
* History of facial paralysis
* Actively receiving treatment related to the temporomandibular joint

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Allodynia | 7 days
  The patients will be evaluated for allodynia with the Allodynia Symptom Checklist. The Allodynia Symptom Checklist include 12 questions about the frequency of various allodynia symptoms in association with headache attacks. Instead of using a dichotomous option (yes or no), the response categories are "never," "rarely," "less than half the time," and "half the time or more." In addition, subjects can also indicate that an item "does not apply to me." That option is used by someone who never shaved their face or someone who never wore a ponytail.
Health-Related Quality | 7 days
  The patients will be evaluated for the quality of life with The Short Form-36. This form is composed of 36 items and eight subscales to evaluate quality of life (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health). The scores of the subscales range between 0 and 100, and higher scores indicate higher quality of life.
Headache-related disability | 3 months
  The patients will be evaluated for headache-related disability with The Migraine Disability Assessment Test. Migraine Disability Assessment scores (numerical scores represent number of days patients missed or lost productivity at work or school, as well as missed days from family/social/leisure activities, and range from little or no disability (0-5) to severe disability (>20).
The impact of headache on quality of life | 3 months
  The patients will be evaluated for the impact of headache on quality of life with 6-item short-form Headache Impact Test. This test is a patient-reported outcome measure used to measure the impact and effect of headache on the ability to function normally in daily life. It consists of 6 questions, total scores may range from 36 to 78 and higher scores reflecting greater impact.
Sleep quality | 7 days
  The patients will be evaluated for sleep quality with the Pittsburgh Sleep Quality Index. It contains 19 self-reported items and 5 items to be completed by a bed partner or roommate, if possible. Scores range from 0 to 3, and are summed to obtain a global score, which ranges from 0 to 21. Higher scores indicate greater sleep disturbance.
Temporomandibular dysfunction | 7 days
  The patients will be evaluated for temporomandibular dysfunction with Helkimo Clinical Dysfunction Index. This index include the following signs: impaired range of movement of the mandible, impaired function of the joint, pain with movement of the mandible, muscle pain, and joint pain. Patients are given a score of 0 points for absence of symptoms, 1 point for mild pain or dysfunction, and 5 points for severe pain or dysfunction.

SECONDARY OUTCOMES:
Descriptive information | 3 days
  Patient's date of birth, gender, education level, body mass index, occupation, marital status, socioeconomic status, age of onset of migraine complaints, descriptive information about migraine attacks (type (with or without aura), duration of attacks, average number of days with pain, severity of pain , companions) will be questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Uğur Uygunoğlu, MD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University- Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No